CLINICAL TRIAL: NCT05595083
Title: Intranasal Dexmedetomidine Versus Intravenous Dexmedetomidine for Improving Quality of the Operative Field in Functional Endoscopic Sinus Surgery: A Randomized Triple-Blind Trial
Brief Title: Intranasal vs. IV Dexmedetomidine in Endoscopic Sinus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed Fouad Algyar, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MKSU 50-9-20
Record Dates: First submitted 2022-10-22; First posted 2022-10-26 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Functional Endoscopic Sinus Surgery; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intranasal dexmedetomidine group (Experimental): patients will receive 1.5 ug/kg intranasal dexmedetomidine diluted with saline + infusion saline
  Interventions: Drug: intranasal dexmedetomidine group
- intravenous dexmedetomidine group (Experimental): patients will receive 0.1- 0.4 ug/kg intravenous infusion dexmedetomidine + intranasal saline.
  Interventions: Drug: intravouns dexmedetomidine group

INTERVENTIONS:
Drug: intranasal dexmedetomidine group — patients will receive 1.5 ug/kg intranasal dexmedetomidine diluted with saline + infusion saline
  Arms: intranasal dexmedetomidine group
Drug: intravouns dexmedetomidine group — patients will receive 0.1- 0.4 ug/kg intravenous infusion dexmedetomidine + intranasal saline.
  Arms: intravenous dexmedetomidine group

SUMMARY:
The aim of this study is to compare intranasal dexmedetomidine versus intravenous dexmedetomidine for improving the quality of the operative field in Functional endoscopic sinus surgery (FESS).

DETAILED DESCRIPTION:
Functional endoscopic sinus surgery (FESS) is a well-established therapeutic option for intractable Cytokine release syndrome (CRS) and other indications. Functional endoscopic sinus surgery (FESS) is a minimally invasive procedure and is commonly performed under controlled hypotensive anesthesia. In case of major bleeding, the risk of complications such as meningitis, blindness, intracranial injury, cerebrospinal fluid [CSF] leakage, and the duration of surgery increase . Intraoperative bleeding is the most common factor that diminishes visibility, resulting in an increased incidence of complications .

Increased bleeding sometimes causes surgeries to end before the due time. Improvement of intraoperative visibility while reducing bleeding is an important task for anesthesiologists during Functional endoscopic sinus surgery (FESS).

For this purpose, several pharmaceuticals have been used successfully to produce controlled hypotension during general anesthesia, for example inhalational anesthetics, direct vasodilators (sodium nitroprusside and nitroglycerin), beta adrenergic antagonists (propranolol and esmolol), alpha adrenergic agonists (clonidine and dexmedetomidine), calcium channel blockers, prostaglandin E1 (alprostadil) and adenosine and l-receptors agonists (remifentanil) .

Dexmedetomidine is a highly selective α2 adreno-receptor agonist with higher affinity to a2 adreno-receptor than clonidine, and this makes dexmedetomidine primarily sedative and anxiolytic .The elimination half-life of dexmedetomidine (t1/2b) is 2 h and the redistribution half-life (t1/2a) is 6 min, and this short half-life makes it an ideal drug for intravenous titration. Potentially desirable effects include decreased requirements for other anesthetics and analgesics. The most common adverse effects associated with Dexmedetomidine include hypotension, bradycardia, and even hypertension.

Intranasal Dexmedetomidine is convenient, effective, and noninvasive and also has useful analgesic and sedative effects in surgical procedures. Cheung's research has shown that intranasal Dexmedetomidine 1 and 1.5 ug/kg in surgical procedures produced significant sedation and less postoperative pain. Several previous research were determined the effect of intranasal dexmedetomidine in several clinical evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Both genders
* American Society of Anesthesiologists (ASA) physical status classification I or II
* Undergoing Functional Endoscopic Sinus Surgery.

Exclusion Criteria:

* Patients with a body mass index > 30 kg/m^2
* contraindications to the use of dexmedetomidine
* history or presence of a significant disease
* significant cardiovascular disease risk factors
* significant coronary artery disease or any known genetic predisposition
* history of any kind of drug allergy
* drug abuse
* psychological or other emotional problems
* special diet or lifestyle
* clinically significant abnormal findings in physical examination
* electrocardiographic (ECG) or laboratory screening
* known systemic disease requiring the use of anticoagulants
* patients with a history of previous Functional Endoscopic Sinus Surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Formmer's scores of surgical field quality | Intraoperatively
  Formmer's scores (a 6-point scale) of surgical field quality will be used to record the amount of bleeding (0= no bleeding; 1= bleeding, so mild it was not even a surgical nuisance; 2= moderate bleeding, a nuisance but without interference; 3= moderate bleeding that moderately compromised surgical; 4= bleeding, heavy but controllable, that significantly interfered; 5= massive uncontrollable bleeding)

SECONDARY OUTCOMES:
Hemodynamics effects | at baseline and every 5 min till the end of procedure
  Heart rate will be recorded
Hemodynamics effects | at baseline and every 5 min till the end of procedure
  Mean arterial blood pressure will be recorded
Pain level | 24 hour postoperatively
  Pain level will be evaluated using numeric rating analogue scale (NRS), which ranges from 0 to 10 points, with 0 indicating no pain, 1-3 indicating mild pain, 4-6 indicating moderate pain, and 7-10 indicating severe pain.
Adverse reactions | 24 hour postoperatively
  Adverse reactions of hemostatic stuffing after Functional endoscopic sinus surgery (FESS) will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Fouad Algyar, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be provided under a reasonable request from the corresponding author.
Supporting Information: Study Protocol
Time Frame: One year after the end of the study